CLINICAL TRIAL: NCT02893462
Title: Setting up a Warehouse of Physiological Data and Biomedical Signals in Adult Intensive Care
Acronym: REASTOC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: REASTOC
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Critical Illness
Keywords: data warehousing; data aggregation; data mining
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is the establishment of a warehouse physiological data and biomedical signal in intensive care adult patients in acute situations from particular records from the Philips Intellivue MP70 monitor.

DETAILED DESCRIPTION:
Cardiopulmonary failures are major public health concerns, due to the aging population. Each of these situations is burdened with a poor prognosis in the medium term and a source of prolonged hospitalizations, generating significant health costs. Early detection and prediction of organ failure could reduce health costs and risks for the patient, offering a reaction early and appropriate medical technology. The proposed approach aims to optimize the knowledge of a complex physiological domain and multi-system, while promoting the automatic transfer of knowledge. The approach proposed data-mining and development of algorithms for detecting and / or predicting a strong potential for disruption because it proposes to apply innovative automated analysis procedures to a fragile patient population, and then a transfer to the medical device industry.

From communicating tools of recording of the signals, the investigator envisage in a global way:

1. the constitution of a warehouse of physiological data of grown-up patients in acute situation (intensive care unit);
2. the development by data mining of a system of detection of organs failures or adverse events basing itself on the application of innovative algorithms, allowing the decision-making operational, from the fusion of arisen ill-assorted events;
3. the use of intelligent tools of auto-learning and elaboration of complex multimodal models for purposes of prediction of events;

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient admitted in Brest University Hospital's intensive care unit for monitoring of vital failure

Exclusion Criteria:

* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of patients admitted in the intensive care unit for monitoring of vital failure
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with physiological signal abnormality | from two to twenty-four hours
  Whereas this is a data mining process (non-deterministic approach), no description can be provided

CONTACTS AND LOCATIONS:
Overall Officials: Erwan L'Her, Professor, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
Ananymized warehouse platform will be shared to other researchers all over the world

REFERENCES:
- [Derived] Bodenes L, N'Guyen QT, Le Mao R, Ferriere N, Pateau V, Lellouche F, L'Her E. Early heart rate variability evaluation enables to predict ICU patients' outcome. Sci Rep. 2022 Feb 15;12(1):2498. doi: 10.1038/s41598-022-06301-9. PMID 35169170
- [Derived] L'Her E, Nazir S, Pateau V, Visvikis D. Accuracy of noncontact surface imaging for tidal volume and respiratory rate measurements in the ICU. J Clin Monit Comput. 2022 Jun;36(3):775-783. doi: 10.1007/s10877-021-00708-x. Epub 2021 Apr 22. PMID 33886075
- [Derived] L'Her E, N'Guyen QT, Pateau V, Bodenes L, Lellouche F. Photoplethysmographic determination of the respiratory rate in acutely ill patients: validation of a new algorithm and implementation into a biomedical device. Ann Intensive Care. 2019 Jan 21;9(1):11. doi: 10.1186/s13613-019-0485-z. PMID 30666472